CLINICAL TRIAL: NCT02961803
Title: MD1003 in Adrenomyeloneuropathy : a Randomized Double Blind Placebo Controlled Study
Brief Title: MD1003-AMN MD1003 in Adrenomyeloneuropathy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: MedDay Pharmaceuticals SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MD1003CT2014-01AMN
Record Dates: First submitted 2016-11-09; First posted 2016-11-11 (Estimated); Last update posted 2017-10-09 (Actual); Status verified 2016-11

CONDITIONS: Adrenomyeloneuropathy; Adrenoleukodystrophy; AMN
Keywords: AMN; MD1003; Adrenomyeloneuropathy; ALD; Adrenoleukodystrophy; Biotin; 2MWT; Two-minute walk test; TW25; Timed 25-Foot Walk
MeSH Terms: conditions — Adrenoleukodystrophy | interventions — Biotin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MD1003 (Experimental): MD1003 100mg capsules, 1 capsule tid for 24 months
  Interventions: Drug: MD1003 100 mg capsule
- Placebo (Placebo Comparator): Placebo capsule, 1 capsule tid for 12 months, then switch to MD1003 100mg capsule, 1 capsule tid for 12 months
  Interventions: Drug: MD1003 100 mg capsule; Drug: Placebo

INTERVENTIONS:
Drug: MD1003 100 mg capsule
  Other Names: High Dose Biotin
Drug: Placebo
  Arms: Placebo

SUMMARY:
The primary objective of the trial is to demonstrate the superiority of biotin at 300 mg/day over placebo in the clinical improvement (walking tests) of patients with adrenomyeloneuropathy

DETAILED DESCRIPTION:
AMN and progressive multiple sclerosis share some similarities including progressive spastic paraparesis and secondary energy failure leading to progressive axonal degeneration. Therefore, it was hypothesized that high doses of biotin might be efficient in patients with AMN.

ELIGIBILITY:
Inclusion Criteria:

* ABCD1 gene mutation identified
* Elevated plasma VLCFA
* Clinical signs of AMN with at least pyramidal signs in the lower limbs and difficulties to walk
* EDSS score ≥ 3.5 and ≤ 6.5
* Normal brain MRI or brain MRI showing :
* abnormalities that can be observed in AMN patients without cerebral demyelination with a maximum Loes score of 4
* and/or stable (≥6 months) cerebral demyelination without gadolinium enhancement with a Loes score ≤12.
* Appropriate steroid replacement if adrenal insufficiency is present
* Likely to be able to participate in all scheduled evaluation visits and complete all required study procedures
* Signed and dated written informed consent to participate in the study in accordance with local regulations
* Affiliated to a Health Insurance

Exclusion Criteria:

* Brain MRI abnormalities with a Loes score > 12 or with gadolinium enhancement
* Any progressive neurological disease other than AMN
* Impossibility to perform the walk tests and the TUG test
* Patients with uncontrolled hepatic disorder, renal or cardiovascular disease, or any progressive malignancy
* Any new medication for AMN including Fampridine initiated less than 1 month prior to inclusion
* Contra-indications for MRI procedure such as subjects with paramagnetic materials in the body, such as aneurysm clips, pacemakers, intraocular metal or cochlear implants.
* Inclusion in another therapeutic clinical trial for ALD
* Not easily contactable by the investigator in case of emergency or not capable to call the investigator

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2014-10; Primary Completion 2016-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Mean change of 2 minutes walking test (2MWT) between Months 12 and baseline | Baseline and 12 Months

SECONDARY OUTCOMES:
Proportion of patients with improved 2-Minutes-Walk-Tests (2MWT) of at least 20% | Baseline, 9 months, 12 months
  at Months 9 and Months 12 compared to the best value among screening and baseline.
Proportion of patients with improved TW25 (time to walk 25 feet) of at least 20% | Baseline, 9 months, 12 months
  at Months 9 and Months 12 compared to the best value among screening and baseline
Mean Change in TW25 (time to walk 25 feet) | Baseline and 12 months
Timed up and Go test (TUG) | 12 Months
Euroqol EQ-5D questionnaire | 12 months
  Quality of Life questionnaire
Qualiveen Questionnaire | 12 Months
  Qualiveen to evaluate urinary function

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Aubourg, MD, Principal Investigator — Hopital Le Kremlin-Bicêtre; Frederic Sedel, MD, Study Director — Medday Pharmeuticals
Locations (4):
- France (2):
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Groupe Hospitalier Pitié-Salpêtrière, Paris
- MS-Ambulanz Fachkrankenhaus Hubertusburg, Wermsdorf, Germany
- Hospital Duran i Reynals / Bellvitge, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No